CLINICAL TRIAL: NCT00917566
Title: Evaluation of Airtraq in Pediatric Population: A Prospective Randomized Study
Brief Title: Evaluation of Airtraq in Pediatric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Khaled Eye Specialist Hospital (Other Government)
Responsible Party: Waleed Riad, King khaled Eye specialist hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP 0909
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Intubation
Keywords: Airtraq; Pediatric

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Airtraq group (Active Comparator): Use Airtraq for intubation
  Interventions: Device: Airtraq
- Macintoch gorup (Active Comparator): Use Macintoch laryngoscope for intubation
  Interventions: Device: Macintoch

INTERVENTIONS:
Device: Airtraq — intubation with airtraq
  Other Names: Optical laryngoscope
  Arms: Airtraq group
Device: Macintoch — use Macintoch laryngoscope for intubation
  Other Names: Standard laryngoscope
  Arms: Macintoch gorup

SUMMARY:
This study indented to evaluate the use of Optical laryngoscope in pediatric

DETAILED DESCRIPTION:
The authors are welling to study how intubation will differ if Airtraq optical laryngoscope used in pediatrics

ELIGIBILITY:
Inclusion Criteria:

* Healthy children undergoing general anesthesia required tracheal intubation.

Exclusion Criteria:

* History of difficult intubation.
* Risk of aspiration.
* Children with cardiovascular disease.
* Children with respiratory disease.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Duration of intubation | two minutes

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Riad, MD, AB, SB, Principal Investigator — King Khaled Eye Specialist Hospital
Locations (1):
- king Khaled Eye Specialist hospital, Riyadh, Riyadh Region, Saudi Arabia